CLINICAL TRIAL: NCT06571877
Title: Impact of Energy Density on Energy Intake During Short- and Long-term Head-down Tilt Bed Rest in Healthy Participants
Brief Title: Impact of Energy Density on Energy Intake During Bed Rest
Acronym: ED-REST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Principal Investigator, Dr. Isabelle Mack, Section Head for Nutrition and Weight Regulation, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 50WB2426A
Record Dates: First submitted 2024-08-15; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Bed Rest; Space Analogue
Keywords: energy intake; energy density; satiety
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: This is a repeated measures randomized controlled cross-over design with an additional randomization on block:
  1) Randomized controlled cross-over experiments are conducted at the end of the first week of the bedrest (days 6-8) and at the end of the bed rest (days 51-53). In total, every participant is tested on 4 days, receiving either the control test meal or the meal with increased fat content in a 1000 ml bowl. 2) Additionally, the 4 campaigns are randomized on block so that either the breakfast or the lunch will be manipulated.
Who Masked: Participant, Outcomes Assessor
Masking Description: The meals are adjusted in energy density without noticeable changes in appearance or taste. These meals have identical ingredients, but the macronutrient proportions are modified. It can be not ruled out that some participants may recognize differences of the meals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control energy density condition (Experimental): Each participant is its own control (cross-over design). Participants receive a bowl with 1000 ml food content consisting of oats, apple pie, grated nuts and milk having an energy density of 1,42 kcal/g. The participants are allowed to eat ad libitum for 45 minutes.
  Interventions: Other: Dietary intervention with manipulation of the energy density
- High energy density condition (Experimental): Participants receive a bowl with 1000 ml food content consisting of oats, apple pie, grated nuts, milk and neutral-tasting vegetable oil having an energy density of 1,84 kcal/g.The participants are allowed to eat ad libitum for 45 minutes.
  Interventions: Other: Dietary intervention with manipulation of the energy density

INTERVENTIONS:
Other: Dietary intervention with manipulation of the energy density — Dietary intervention with manipulation of the energy density either during breakfast or during lunch

SUMMARY:
Brief summary: This study is conducted in the context of a 60 days strict bed-rest study with 6° head-down-tilt (HDT) body position. Food intake can be challenging during bed-rest due to loss of appetite and constantly feeling full. The study aims to assess whether or not energy intake varies during a meal when the energy density of a meal is increased by the fat content. This experiment follows a crossover design with repeated measures within subjects. The order of experimental conditions is balanced among participants and sex, and the assignment of orders to participants is randomly. On each test day, participants are provided with breakfast, lunch, and dinner as usual. Across test days, the ED of breakfast (24 participants) or lunch (24 participants) is modified to two levels: the standard level and an increased level (+ 0.42 kcal/g compared to the standard). The meals are adjusted in energy density without noticeable changes in appearance or taste. These meals have identical ingredients, but the macronutrient proportions are modified. Entrées with increased fat content are prepared by incorporating neutral-tasting vegetable oil into the standard recipes. Participants receive their meals and are given the flexibility to eat ad libitum for 45 minutes. To comply with the strict bed rest rules, the next meal will be used for counterbalancing total energy intake over the day if necessary. In case of problems, a nutrient drink could be used to assure the requested total energy intake in order to maintain body weight.The experiments are conducted during 4 campaigns, each campaign consisting of 12 participants.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally healthy test subjects that declare their willingness to participate in the entire study and successfully pass the psychological and medical screening
* Aged between 24 and 55 years
* Body mass index between 18 to 28 kg/m2
* Body height between 153 to 190 cm (+/- 2 cm)
* Signed informed consent
* Demonstrable medical insurance and official certificate of absence of criminal record
* No less than 2 SD below the average normal bone mineral density (measured by dual-energy x-ray absorptiometry) for hip and lumbar spine (i.e., mean peak bone mineral density of Caucasian, sex-matched young adults) denoted by T-score (T-score > -2)
* Demonstrable dentist certificate
* Hormonal contraception for female participants is allowed, but details (manufacturer, doses, dates) must be reported

Exclusion Criteria:

Candidate subject exclusion criteria for the study will include the following:

* Any infectious, genetic, autoimmune, endocrinological, hematological, cardiovascular, lung, gastroenterological, kidney, rheumatic, muscle, bone, orthopedic, dermatological, gynecological, urological, ophthalmological, otorhinolaryngological, neurological or psychiatric disease (see at the end of document; a) that precludes a safe participation in the study or might significantly impact scientific results of the study according to the study physician
* Drug, medication or alcohol abuse (regular consumption of more than 30 g alcohol/day)
* Smoker within 6 months prior to enrollment
* Any long-term medication use that might significantly impact scientific results of the study (for instance bisphosphonate therapy, anti-hypertensives, gastro-esophageal reflux).

Special dietary requests, that cannot be provided by the project team (e.g. vegan, vegetarian or other ineligible diet)

* Claustrophobia
* Increased intraocular pressure
* Hyperopia / Myopia > +/- 5.0 Diopters
* Astigmatism > 3 Diopters
* History of laser surgery of the eye, glaucoma and retinal surgery
* Any ocular condition that would significantly impact visual function
* Significant chronic gastro-esophageal reflux precluding a safe participation in the study
* Clinically relevant allergy (e.g. requirement to carry a stand-by emergency injection), that precludes a safe participation in the study
* History of chronic back complaints, that precludes a safe participation in the study
* History of kidney stones
* Anemia: Hemoglobin under normal values (see at the end of document; b). (Normal values of Hemoglobin for men: 13.0-17.5 g/dl; women 12.0-16.0 g/dl)
* Elevated risk of thrombosis (see at the end of document; c)
* Inability to successfully complete a 10-minute upright posture test without clinically relevant orthostatic symptoms
* Current or history of hemorrhagic diathesis or coagulations disorders
* History of spinal cord disease, including radiculopathy, myelopathy, or neuropathy
* History of disorders affecting CSF circulation (i.e. hydrocephalus, idiopathic intracranial hypertension) History of more than one depressive episode and/or history of a severe depressive episode, such as requiring inpatient or intensive outpatient treatment
* Known chronic tinnitus
* Hearing loss (bi-lateral or one-sided) precluding successful participation in the study
* Female candidate is pregnant or breast-feeding
* Female candidate is in menopause or post-menopause, unless on hormone replacement therapy (but not treated with bisphosphonates or anti-resorptives)
* Female candidate stopped hormonal contraception medication up to 3 months prior to study start
* Metal implants (or objects like metallic slivers in the eyes, or bullets or shrapnel in the body) or other kinds of bone synthesis materials, implanted medical devices, tattoos or permanent make-up incompatible with MRI
* Participation in a (clinical) study within the last 3 months before start of this study that significantly confounds participation in the study Any other condition which makes the test subject unsuitable for study inclusion in the opinion of the project team

Explanations to exclusion criteria (a-c)

1. History of single episode of prolonged grief or mild depression with no symptoms in the 12 months prior to study start is acceptable
2. Normal values from: https://www.lab-quade.de/leistungen/?idLoc=1
3. A thrombosis risk stratification will be conducted according to clinical standards: in the anamnesis, the subject will be extensively questioned for thrombosis risk factors and assessed by means of specific analytical laboratory methods for assessing thrombosis risk using thrombophilia screening

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-24 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy intake in kcal | Measurments taken at days 6, 8, 51 and 53 in the 60 days head down tilt period.
  Energy intake is calculated by measuring the amount of food before and after the experiment and precalculation of the energy content of the meals

SECONDARY OUTCOMES:
Amount of food intake in g | Measurments taken at days 6, 8, 51 and 53 in the 60 days head down tilt period.
  The amount of food intake is calculated by measuring the amount of food before and after the experiment
Composite appetite score measured by 10 cm visual analogue scales (VAS) | Measurments taken at days 6, 8, 51 and 53 in the 60 days head down tilt period before the meal, 30 minutes, 45 minutes and 60 minutes after the meal and directly before the next meal (either lunch or dinner)
  Appetite perception is measured using validated 100 mm VAS for hunger, satisfaction, fullness, and prospective food consumption (Flint et al., 2000). The composite score is calculated as follows: ([hunger + prospective food consumption + (100-fullness) + (100-satisfaction)]/4) by Stubbs et al., 2000
Visual analogue scale for perception of portion size | Measurments taken at days 6, 8, 51 and 53 in the 60 days head down tilt period before the meal, 30 minutes, 45 minutes and 60 minutes after the meal and directly before the next meal (either lunch or dinner)
  Portion size is measured using a 100 mm VAS.
Emotional response | Measurments taken at days 6, 8, 51 and 53 in the 60 days head down tilt period before the meal, 30 minutes and 60 minutes after the meal and directly before the next meal (either lunch or dinner)
  Emotional response is used using the Self assessment manikin (Bradley & Lang, 1994)
Number of participants assigned to countermeasures for consequences of long-term bed rest | Allocation to countermeasure test arms is done ahead of the bed rest study, at least 4 weeks ahead bed rest.
  During bed rest, the participants are allocated to 4 arms of different countermeasures for consequences of long-term bed red which is independent of this food study. These countermeasures include: Arm 1: Electrical Muscle Stimulation; Arm 2: Proprioceptive Training; Arm 3: Exercise plus proprioceptive Training; Arm 4: Control.
  This information on "bed rest countermeasure" will be added as a co-variate.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mack, PD Dr., Principal Investigator — Internal Medicine VI, University Hospital Tuebingen, Osianderstr. 5, 72076 Tuebingen, Germany
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No